CLINICAL TRIAL: NCT03144674
Title: A Phase 2, Open-Label, 2-Cohort Study of INCB050465, a PI3Kδ Inhibitor, in Subjects With Relapsed or Refractory Marginal Zone Lymphoma With or Without Prior Exposure to a BTK Inhibitor (CITADEL-204)
Brief Title: A Study of INCB050465 in Subjects With Relapsed or Refractory Marginal Zone Lymphoma (CITADEL-204)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INCB 50465-204 (CITADEL-204); Parsaclisib (Other: Incyte Corporation); 2017-000970-12 (EudraCT Number)
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Results first posted 2022-02-10 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Lymphoma
Keywords: Marginal zone lymphoma; phosphatidylinositol 3-kinase (PI3K)δ inhibitor; indolent (slow-growing) non-Hodgkin lymphoma B-cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, B-Cell, Marginal Zone | interventions — parsaclisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1- Closed to Further enrollment (Experimental): Participants who have received prior ibrutinib.
  Interventions: Drug: Parsaclisib
- Cohort 2 (Experimental): Participants who have not received a prior BTK inhibitor.
  Interventions: Drug: Parsaclisib

INTERVENTIONS:
Drug: Parsaclisib — Parsaclisib at the protocol-defined dose.
  Other Names: INCB050465

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of two parsaclisib treatment regimens in participants diagnosed with relapsed or refractory marginal zone lymphoma (MZL) who are naive to or were previously treated with a Bruton's tyrosine kinase (BTK) inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged 18 or older (except in South Korea, aged 19 or older).
* Histologically confirmed marginal zone lymphoma, including extranodal, nodal, and splenic subtypes.
* Radiographically measurable lymphadenopathy or extranodal lymphoid malignancy (defined as the presence of ≥ 1 lesion that measures > 1.5 cm in the longest transverse diameter and ≥ 1.0 cm in the longest perpendicular diameter.
* Participants with splenic MZL who do not meet the radiographically measurable disease criteria described herein are eligible for participation provided that bone marrow infiltration of MZL is histologically confirmed.
* Participants must be willing to undergo an incisional or excisional lymph node or tissue biopsy or provide a lymph node or tissue biopsy from the most recent available archival tissue.
* Eastern Cooperative Oncology Group performance status 0 to 2.

Exclusion Criteria:

* Evidence of diffuse large B-cell transformation.
* History of central nervous system lymphoma (either primary or metastatic) or leptomeningeal disease.
* Prior treatment with idelalisib, other selective PI3Kδ inhibitors, or a pan-PI3K inhibitor.
* Allogeneic stem cell transplant within the last 6 months, or autologous stem cell transplant within the last 3 months before the date of the first dose of study treatment.
* Active graft versus host disease.
* Subjects positive for hepatitis B surface antigen or hepatitis B core antibody will be eligible if they are negative for HBV-DNA. Subjects positive for anti-HCV antibody will be eligible if they are negative for HCV-RNA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2024-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred Zheng, MD, Study Director — Incyte Corporation
Locations (86):
- United States (33):
  - University of Alabama At Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Arizona Oncology Associates, Tempe, Arizona
  - Torrance Health Association, Redondo Beach, California
  - Sansum Clinic, Santa Barbara, California
  - Central Coast Medical Oncology, Santa Maria, California
  - UCLA Healthcare Hematology-Oncology, Santa Monica, California
  - St. Joseph Heritage Healthcare, Santa Rosa, California
  - Innovative Clinical Research Institute, Whittier, California
  - Loyola University Medical Center, Whittier, California
  - Valley View Hospital, Glenwood Springs, Colorado
  - St. Mary'S Hospital Regional Cancer Center, Grand Junction, Colorado
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Advanced Pharma Cr, Miami, Florida
  - Boca Raton Clinical Research Medical Inc., Plantation, Florida
  - Asclepes Research Centers, Weeki Wachee, Florida
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - Rush University Medical Center - Consultants in Hematology, Chicago, Illinois
  - Clinical Trials of Swla Llc, Lake Charles, Louisiana
  - University of Michigan Cancer Center, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Saint Luke'S Hospital of Kansas City, Kansas City, Missouri
  - COMPREHENSIVE CANCER CeNTERS OF NEVADA - TWAIN, Las Vegas, Nevada
  - Clinical Research Alliance, New Hyde Park, New York
  - Nyu Cancer Institute, New York, New York
  - Hematology Oncology Associates of Rockland, Nyack, New York
  - White Plains Hospital, White Plains, New York
  - Duke University Medical Center, Durham, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Charleston Hematology Oncology Associates Pa, Charleston, South Carolina
  - Renovatio Clinical, The Woodlands, Texas
  - University of Washington - Seattle Cancer Care Alliance, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Aou Maggiore Della Carita, Rosario, Argentina
- Australia (3):
  - Icon Cancer Care, Auchenflower, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Calvary North Adelaide Hospital, North Adelaide, South Australia
- Belgium (3):
  - Cliniques Universitaires Ucl Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Universitaire Ziekenhuis Leuven - Gasthuisberg, Leuven
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Zealand University Hospital, Roskilde
- France (8):
  - Avicenne Hospital, Bobigny
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Chu Limoges - Hospital Le Cluzeau, Limoges
  - Hopital Saint-Louis, Paris
  - H�Pital Universitaire Piti�-Salp�Tri�Re, Paris
  - Hospices Civils de Lyon Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Henri Becquerel, Rouen
  - Institute Gustave Roussy (Igr), Villejuif
- Germany (6):
  - Universit�Tsklinikum Essen, Essen
  - Universitatsmedizin Gottingen, Göttingen
  - Universit�Tsklinikum Schleswig-Holstein, Kiel
  - Klinikum Ludwigshafen, Ludwigshafen
  - Universitatsmedizin Der Johannes Gutenberg-Universitat Mainz Iii, Mainz
  - Universit�Tsklinikum Ulm, Ulm
- Israel (5):
  - Rambam Medical Center, Haifa
  - Hadassah Hebrew University Medical Center Ein Karem Hadassah, Jerusalem
  - Rabin Medical Center - Beilinson Hospital, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (9):
  - University of Bologna, Institute of Haematology �L. E A. Ser�Gnoli�, Bologna
  - Istituto Scientifico Romagnolo Per Lo Studio E La Cura Dei Tumori, Meldola
  - Fondazione Centro San Raffaele - Milano, Milan
  - Fondazione Irccs Istituto Nazionale Dei Tumori, Milan
  - Azienda Ospedaliera San Gerardo Di Monza, Monza
  - Azienda Ospedaliera Ospedali Riuniti "Villa Sofia - Cervello", Palermo
  - Presidio Ospedaliero Pescara, Pescara
  - Ospedale Delle Croci - Ematologia Ravenna, Ravenna
  - Sapienza University, Rome
- Poland (5):
  - Centrum Onkologii-Instytut Im. Marii Sklodowskiej-Curie, Gdansk
  - Szpitale Wojew�Dzkie W Gdyni Sp�?Ka Z Ograniczon? Odpowiedzialno?Ci?, Gdansk
  - Malopolskie Centrum Medyczne S.C., Krakow
  - Klinika Transplantacji Komorel Krwiotworczych, Warsaw
  - Centrum Onkologii-Instytut Im. Marii Sklodowskiej-Curie, Warsaw
- Spain (7):
  - Hospital General Universitari Vall D Hebron, Barcelona
  - Ico Institut Catala D Oncologia, Barcelona
  - Hgu Gregorio Maranon, Madrid
  - Hospital Universitario Hm Sanchinarro, Madrid
  - Hospital Universitario Quironsalud Madrid, Madrid
  - Hospital Puerta de Hierro, Majadahonda
  - Hospital Universitario de Salamanca, Salamanca
- United Kingdom (4):
  - Birmingham Heartlands Hospital, Birmingham
  - Kent Oncology Centre - Maidstone Hospital, Maidstone
  - Norfolk and Norwich University Hospital, Norwich
  - University of Southampton, Southampton

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled participants at 46 study centers in the United States, Italy, Israel, France, Spain, Poland, Belgium, Great Britain, and Germany.
Pre-assignment Details: A total of 110 participants diagnosed with relapsed or refractory marginal zone lymphoma were enrolled into two cohorts based on previous treatment with ibrutinib as Cohort 1: those who were exposed to ibrutinib before enrollment and Cohort 2: those who were not exposed to Bruton's tyrosine kinase (BTK) inhibitor before enrollment. Participants were further allocated to Treatments A and B in each Cohort to receive parsaclisib.
Groups:
- Cohort 1: Treatment A (Exposed to Ibrutinib): Participants received parsaclisib 20 milligrams (mg), orally, once daily (QD) for 8 weeks followed by 20 mg once weekly (QW), for up to 52 weeks. Participants who were exposed to ibrutinib before enrollment were included in this group.
- Cohort 1: Treatment B (Exposed to Ibrutinib): Participants received parsaclisib 20 mg, orally, QD for 8 weeks followed by 2.5 mg QD, for up to 52 weeks. Participants who were exposed to ibrutinib before enrollment were included in this group.
- Cohort 2: Treatment A (Bruton's Tyrosine Kinase Inhibitor Naïve): Participants received parsaclisib 20 mg tablets, orally, QD for 8 weeks followed by 20 mg tablets QW, for up to 52 weeks. Participants who were not exposed to BTK inhibitor before enrollment were included in this group
- Cohort 2: Treatment B (Bruton's Tyrosine Kinase Inhibitor Naïve): Participants received parsaclisib 20 mg tablets, orally, QD for 8 weeks followed by 2.5 mg tablets QD, for up to 52 weeks. Participants who were not exposed to BTK inhibitor before enrollment were included in this group.
Period: Overall Study
Arm/Group | Cohort 1: Treatment A (Exposed to Ibrutinib) | Cohort 1: Treatment B (Exposed to Ibrutinib) | Cohort 2: Treatment A (Bruton's Tyrosine Kinase Inhibitor Naïve) | Cohort 2: Treatment B (Bruton's Tyrosine Kinase Inhibitor Naïve)
Started | 4 | 6 | 28 | 72
Completed | 0 | 2 | 13 | 26
Not Completed | 4 | 4 | 15 | 46
Not completed — Participant Transferred to Rollover Study | 1 | 1 | 5 | 6
Not completed — Death | 3 | 2 | 6 | 24
Not completed — Lost to Follow-up | 0 | 1 | 0 | 4
Not completed — Withdrawal by Participant | 0 | 0 | 2 | 6
Not completed — Discharged from the Trust | 0 | 0 | 1 | 0
Not completed — Exclusion Criteria Met | 0 | 0 | 1 | 0
Not completed — Changed Physicians | 0 | 0 | 0 | 1
Not completed — Removed for Safety | 0 | 0 | 0 | 1
Not completed — Site Closed | 0 | 0 | 0 | 1
Not completed — Histological Criteria Not Met | 0 | 0 | 0 | 1
Not completed — Multifactorial Cognitive Decline | 0 | 0 | 0 | 1
Not completed — Progression of Chronic Lymphocytic Leukemia | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants enrolled in the study who received at least 1 dose of parsaclisib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Treatment A (Exposed to Ibrutinib) | Cohort 1: Treatment B (Exposed to Ibrutinib) | Cohort 2: Treatment A (Bruton's Tyrosine Kinase Inhibitor Naïve) | Cohort 2: Treatment B (Bruton's Tyrosine Kinase Inhibitor Naïve) | Total
Number analyzed (Participants) | 4 | 6 | 28 | 72 | 110
Age, Continuous [Mean (Full Range); unit: years] | 73.5 [71 to 76] | 72.2 [65 to 78] | 68.1 [52 to 86] | 69.8 [35 to 95] | 69.6 [35 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 16 | 31 | 53
  Male | 2 | 2 | 12 | 41 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 3 | 4 | 9
  Not Hispanic or Latino | 3 | 4 | 19 | 57 | 83
  Unknown or Not Reported | 1 | 0 | 6 | 11 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1 | 2
  White | 3 | 5 | 23 | 60 | 91
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 5 | 10 | 16

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Based on Lugano Classification Criteria
Description: ORR=percentage of participants with complete response(CR) or partial response(PR) per revised response criteria for lymphomas,determined by independent review committee(IRC).Criteria for CR:1.Target nodes/nodal masses of lymph nodes,extralymphatic sites regressed to≤1.5cm in longest dimension transverse diameter of lesion(LDi);2.Absence of non-measured lesion;3.Organ enlargement regressed to normal;4.No new lesions;5.Normal bone marrow morphology;if indeterminate,immunohistochemistry negative.Criteria for PR:1.Lymph nodes,extralymphatic sites- ≥50%decrease in sum of product of perpendicular diameters for multiple lesions(SPD)of up to 6 target measurable nodes,extranodal sites;if lesion is too small to measure on computed tomography(CT),assign 5mm×5mm as default;if no longer visible,0×0mm.Node >5mm×5mm but smaller than normal,use actual measurement.2.Absent/regressed non-measured lesions,no increase.3.Organ enlargement-Spleen regressed by >50%in length beyond normal.4.No new lesions.
Time Frame: Up to approximately 161 weeks
Population: Full Analysis Set: all participants enrolled in the study who received at least 1 dose of parsaclisib
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Treatment A (Exposed to Ibrutinib) | Cohort 1: Treatment B (Exposed to Ibrutinib) | Cohort 2: Treatment A (Bruton's Tyrosine Kinase Inhibitor Naïve) | Cohort 2: Treatment B (Bruton's Tyrosine Kinase Inhibitor Naïve)
Number analyzed (Participants) | 4 | 6 | 28 | 72
percentage of participants | 50.0 [6.8 to 93.2] | 33.3 [4.3 to 77.7] | 57.1 [37.2 to 75.5] | 58.3 [46.1 to 69.8]

2. Secondary Outcome: Duration of Response (DOR)
Description: DOR=time from first documented evidence of CR or PR until disease progression or death from any cause among participants who achieve an objective response as determined by IRC. Criteria for CR: 1.Target nodes/nodal masses of lymph nodes and extralymphatic sites must regress to ≤ 1.5 cm in LDi; 2. Absence of non-measured lesion; 3.Organ enlargement regressed to normal; 4.No new lesions; 5.Bone marrow must be normal by morphology; if indeterminate, immunohistochemistry negative. The criteria for PR included: 1.Lymph nodes and extralymphatic sites- a. ≥50% decrease in SPD of up to 6 target measurable nodes and extranodal sites; b. when a lesion is too small to measure on CT, assign 5 mm×5 mm as the default; c.when no longer visible, 0×0 mm. For a node >5 mm×5 mm but smaller than normal, use actual measurement. 2.Non-measured lesions- Absent/regressed, but no increase. 3. Organ enlargement-Spleen must have regressed by >50% in length beyond normal. 4.No new lesions.
Time Frame: Up to 1305 days
Population: Full Analysis Set: all participants enrolled in the study who received at least 1 dose of parsaclisib. Only participants with objective response were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Treatment A (Exposed to Ibrutinib) | Cohort 1: Treatment B (Exposed to Ibrutinib) | Cohort 2: Treatment A (Bruton's Tyrosine Kinase Inhibitor Naïve) | Cohort 2: Treatment B (Bruton's Tyrosine Kinase Inhibitor Naïve)
Number analyzed (Participants) | 2 | 2 | 17 | 41
months | NA [NA to NA] — The median and lower and upper limits of the 95% confidence interval (CI) were not estimable due to the low number of participants with events of response. | NA [NA to NA] — The median and lower and upper limits of the 95% CI were not estimable due to the low number of participants with events of response. | 16.69 [3.71 to NA] — The upper limit of the 95% CI was not estimable due to the low number of participants with events of response. | 13.57 [8.05 to 17.74]

3. Secondary Outcome: Complete Response Rate (CRR) Based on Lugano Classification Criteria
Description: CRR is defined as the percentage of participants with a CR as determined by an IRC. The criteria for CR included: 1.Target nodes/nodal masses of lymph nodes and extralymphatic sites must regress to ≤ 1.5 cm in LDi; 2. Absence of non-measured lesion; 3.Organ enlargement regressed to normal; 4.No new lesions; 5.Bone marrow must be normal by morphology; if indeterminate, immunohistochemistry negative.
Time Frame: Up to 1305 days
Population: Full Analysis Set: all participants enrolled in the study who received at least 1 dose of parsaclisib
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Treatment A (Exposed to Ibrutinib) | Cohort 1: Treatment B (Exposed to Ibrutinib) | Cohort 2: Treatment A (Bruton's Tyrosine Kinase Inhibitor Naïve) | Cohort 2: Treatment B (Bruton's Tyrosine Kinase Inhibitor Naïve)
Number analyzed (Participants) | 4 | 6 | 28 | 72
percentage of participants | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 45.9] | 10.7 [2.3 to 28.2] | 4.2 [0.9 to 11.7]

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from the date of the first dose of study treatment until the earliest date of disease progression, as determined by radiographic disease assessment provided by an IRC, or death from any cause.
Time Frame: Up to 1305 days
Population: Full Analysis Set: all participants enrolled in the study who received at least 1 dose of parsaclisib
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Treatment A (Exposed to Ibrutinib) | Cohort 1: Treatment B (Exposed to Ibrutinib) | Cohort 2: Treatment A (Bruton's Tyrosine Kinase Inhibitor Naïve) | Cohort 2: Treatment B (Bruton's Tyrosine Kinase Inhibitor Naïve)
Number analyzed (Participants) | 4 | 6 | 28 | 72
months | NA [NA to NA] — The median and lower and upper limits of the 95% CI were not estimable due to the low number of participants with events. | NA [NA to NA] — The median and lower and upper limits of the 95% CI were not estimable due to the low number of participants with events. | 19.42 [8.77 to NA] — The upper limit of the 95% CI was not estimable due to the low number of participants with events. | 17.74 [11.53 to 22.34]

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of the first dose of study treatment until death from any cause.
Time Frame: Up to 2354 days
Population: Full Analysis Set: all participants enrolled in the study who received at least 1 dose of parsaclisib
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Treatment A (Exposed to Ibrutinib) | Cohort 1: Treatment B (Exposed to Ibrutinib) | Cohort 2: Treatment A (Bruton's Tyrosine Kinase Inhibitor Naïve) | Cohort 2: Treatment B (Bruton's Tyrosine Kinase Inhibitor Naïve)
Number analyzed (Participants) | 4 | 6 | 28 | 72
months | 18.94 [7.26 to NA] — The upper limit of the 95% CI was not estimable due to the low number of participants with events. | NA [3.22 to NA] — The median was not reached and the upper limit of the 95% CI was not estimable due to the low number of participants with events. | NA [59.60 to NA] — The median was not reached and the upper limit of the 95% CI was not estimable due to the low number of participants with events. | 63.54 [39.72 to NA] — The median was not reached and the upper limit of the 95% CI was not estimable due to the low number of participants with events.

6. Secondary Outcome: Best Percent Change From Baseline in Target Lesion Size
Description: Target lesion size is measured by the sum of the product of diameters of all target lesion sizes and is determined by the IRC. The best percent change from Baseline is defined as the largest decrease, or smallest increase (if no decrease available), from Baseline in target lesion sizes on/before new (next-line) anti-lymphoma therapy during the study. Baseline is the last nonmissing measurement obtained before the first administration of study drug. A negative percent change from Baseline indicates improvement.
Time Frame: Up to 1305 days
Population: Full Analysis Set: all participants enrolled in the study who received at least 1 dose of parsaclisib. The overall number of participants analyzed is the number of participants with splenomegaly and data available for analysis.
Measure: Mean (Standard Deviation); unit: percent change in lesion size
Groups:
- Cohort 2: Bruton's Tyrosine Kinase Inhibitor Naïve (Treatment A): Participants received parsaclisib 20 mg tablets, orally, QD for 8 weeks followed by 20 mg tablets QW, for up to 52 weeks. Participants who were not exposed to BTK inhibitor before enrollment were included in this group.
- Cohort 2: Bruton's Tyrosine Kinase Inhibitor Naïve (Treatment B): Participants received parsaclisib 20 mg tablets, orally, QD for 8 weeks followed by 2.5 mg tablets QD, for up to 52 weeks. Participants who were not exposed to BTK inhibitor before enrollment were included in this group.
Arm/Group | Cohort 1: Treatment A (Exposed to Ibrutinib) | Cohort 1: Treatment B (Exposed to Ibrutinib) | Cohort 2: Bruton's Tyrosine Kinase Inhibitor Naïve (Treatment A) | Cohort 2: Bruton's Tyrosine Kinase Inhibitor Naïve (Treatment B)
Number analyzed (Participants) | 4 | 5 | 20 | 51
percent change in lesion size | -48.83 (21.193) | -54.84 (21.454) | -71.22 (18.566) | -66.76 (19.971)

7. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence associated with use of a drug in humans, whether or not considered drug related, that occurs after a participant provides informed consent. A TEAE is any AE either reported for the first time or worsening of a pre-existing event after first dose of study drug and within 30 days of the last administration of study drug regardless of starting new anti-lymphoma therapy. A SAE is any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, leads to a congenital anomaly/birth defect or is considered to be an important medical event that may not result in death, be immediately life-threatening, or require hospitalization but may be considered serious when, based on appropriate medical judgment, the event may jeopardize the participant or may require medical or surgical intervention.
Time Frame: From first dose of study drug up to 1980 days
Population: Safety Population: all enrolled participants who received at least 1 dose of parsaclisib
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Treatment A (Exposed to Ibrutinib) | Cohort 1: Treatment B (Exposed to Ibrutinib) | Cohort 2: Treatment A (Bruton's Tyrosine Kinase Inhibitor Naïve) | Cohort 2: Treatment B (Bruton's Tyrosine Kinase Inhibitor Naïve)
Number analyzed (Participants) | 4 | 6 | 28 | 72
percentage of participants
  TEAEs | 100.0 | 83.3 | 92.9 | 97.2
  SAEs | 50.0 | 33.3 | 32.1 | 63.9

ADVERSE EVENTS:
Time Frame: up to 2354 days
Description: Adverse events have been reported for members of the Safety Population, comprised of all enrolled participants who received at least 1 dose of parsaclisib.
Arm/Group | Cohort 1: Treatment A (Exposed to Ibrutinib) | Cohort 1: Treatment B (Exposed to Ibrutinib) | Cohort 2: Treatment A (Bruton's Tyrosine Kinase Inhibitor Naïve) | Cohort 2: Treatment B (Bruton's Tyrosine Kinase Inhibitor Naïve)
All-Cause Mortality (participants affected / at risk) | 3/4 | 2/6 | 6/28 | 25/72
Serious Adverse Events (participants affected / at risk) | 2/4 | 2/6 | 9/28 | 46/72
Other Adverse Events (participants affected / at risk) | 4/4 | 5/6 | 25/28 | 67/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Treatment A (Exposed to Ibrutinib) (N=4) | Cohort 1: Treatment B (Exposed to Ibrutinib) (N=6) | Cohort 2: Treatment A (Bruton's Tyrosine Kinase Inhibitor Naïve) (N=28) | Cohort 2: Treatment B (Bruton's Tyrosine Kinase Inhibitor Naïve) (N=72)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Blood calcium increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Cytomegalovirus colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus infection reactivation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterobacter sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Faecal volume increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (5)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal infarction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Marginal zone lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Microangiopathic haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oliguria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 2 (3) | 7 (8)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Yersinia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Treatment A (Exposed to Ibrutinib) (N=4) | Cohort 1: Treatment B (Exposed to Ibrutinib) (N=6) | Cohort 2: Treatment A (Bruton's Tyrosine Kinase Inhibitor Naïve) (N=28) | Cohort 2: Treatment B (Bruton's Tyrosine Kinase Inhibitor Naïve) (N=72)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 10 (11)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (5) | 7 (11)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 4 (5) | 10 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 4 (4) | 9 (11)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (6) | 6 (9)
Asthenia (General disorders) | 0 (0) | 0 (0) | 4 (6) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 4 (5)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 2 (3)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
COVID-19 (Infections and infestations) | 1 (2) | 0 (0) | 4 (4) | 4 (4)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (6)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (5) | 11 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 5 (8) | 22 (24)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (3) | 11 (12)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (3) | 9 (19) | 37 (66)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 9 (11)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 7 (7)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 2 (2) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (3) | 3 (9)
Fatigue (General disorders) | 1 (1) | 1 (1) | 3 (5) | 11 (11)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 10 (12)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 4 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (8)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 6 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (11)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Infected bite (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 2 (4) | 3 (4)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (4) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (3) | 4 (4)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 4 (4) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 13 (18)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 4 (5) | 10 (20)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (2) | 2 (7) | 4 (9)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 3 (3) | 9 (9)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (3) | 3 (4)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 4 (11)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 5 (6) | 11 (13)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (2) | 4 (8) | 10 (14)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 5 (8) | 11 (12)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 5 (6)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (6) | 5 (5)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (4) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 11 (13)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 6 (9)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (5) | 5 (8)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (4)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2019-12-23): https://cdn.clinicaltrials.gov/large-docs/74/NCT03144674/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/74/NCT03144674/SAP_001.pdf